CLINICAL TRIAL: NCT06841770
Title: Delivery of Oligodendrocyte Progenitor Cells for Spinal Cord Injury: Evaluation of a Novel Device (DOSED)
Brief Title: A Study to Evaluate the Safety of a Delivery Device for Administering LCTOPC1 in Participants With Spinal Cord Injury
Acronym: DOSED
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Lineage Cell Therapeutics, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: LCTOPC1-SCI-03
Record Dates: First submitted 2025-02-11; First posted 2025-02-24 (Actual); Last update posted 2026-02-12 (Actual); Status verified 2026-02

CONDITIONS: Spinal Cord Injury Cervical; Spinal Cord Injury Thoracic; Spinal Cord Injury, Acute; Spinal Cord Injury; Spinal Cord Injury, Chronic
Keywords: Spinal Cord Injury; DOSED; Subacute spinal cord injury; Oligodendrocyte Progenitor Cell; Chronic spinal cord injury; Stem Cell Transplant; Cervical spinal cord injury; Thoracic spinal cord injury; Paralysis; Quadriplegia; Tetraplegia
MeSH Terms: conditions — Spinal Cord Injuries; Bronchiolitis Obliterans Syndrome; Paralysis; Quadriplegia

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- LCTOPC1 (Experimental): Open Label Single Injection of LCTOPC1 at a Single Time Point
  Interventions: Biological: OPC1

INTERVENTIONS:
Biological: OPC1 — One injection of 10 million LCTOPC1 cells will be delivered to the target injection site of the damaged spinal tissue.

SUMMARY:
The DOSED clinical study evaluates the safety and utility of a novel delivery device to deliver LCTOPC1, a cell therapy, to the spinal cord of patients with a spinal cord injury (SCI). LCTOPC1 is designed to replace or support cells that are absent or dysfunctional due to traumatic injury, with a goal to help improve the quality of life and restore or augment functional activity in persons suffering from a traumatic cervical or thoracic injuries.

DETAILED DESCRIPTION:
LCTOPC1-SCI-03 DOSED study is a Phase 1b, open-label, multi-center, device safety study designed to assess the safety of a novel delivery device for administering a one-time injection of LCTOPC1. The study will enroll 3-5 participants with subacute (21 to 42 days post-injury) spinal cord injuries and 3-5 participants with chronic (1 to 5 years post-injury) spinal cord injuries. Eligible participants must have either sensorimotor complete (AIS-A) or motor complete / sensory incomplete spinal cord injuries (AIS-B), located in the cervical (C4-C7) or thoracic (T1-T10) regions. The first four patients will be enrolled sequentially subsequent to meeting safety requirements. Participants will be monitored for long-term safety for up to 10 years following the administration of LCTOPC1.

ELIGIBILITY:
Inclusion Criteria:

1. Sensorimotor complete, traumatic SCI (ASIA Impairment Scale A) or sensory incomplete, traumatic SCI (ASIA Impairment Scale B)
2. For subjects with subacute injury, International Standards for Neurological Classification of SCI (ISNCSCI) Neurological Level of Injury (NLI) from C-4 to T-10 occurring 21 to 42 days prior to LCTOPC1 injection
3. For subjects with chronic injury, ISNCSCI NLI from C-4 to T-10 and more than 30 days without clinical improvement from last assessment, occurring 1 to 5 years prior to LCTOPC1 injection
4. Individuals must have at least one upper extremity ISNCSCI key muscle with at least 1/5 strength
5. 18 through 65 years of age, inclusive, at time of consent
6. Single injury with sufficient visualization of the spinal cord injury epicenter and lesion margins to enable post-injection safety monitoring
7. Informed consent for this protocol must be provided and documented (i.e., signed ICF)
8. Able to participate in an elective surgical procedure to inject LCTOPC1 21 days or later following SCI
9. Female subjects of child-bearing potential must agree to the use of contraception for 1 year following LCTOPC1 injection; male subjects must agree to use contraception to prevent pregnancy in any female partners of child-bearing potential for 1 year following LCTOPC1 injection

Exclusion Criteria:

1. SCI due to penetrating trauma
2. Traumatic anatomical transection, laceration, or inadequate decompression of the spinal cord based on prior surgery or MRI
3. Any concomitant injury that interferes with the performance, interpretation, or validity of neurological examinations, such as multiple spinal cord lesions, brachial/lumbar plexus injury, cauda equina injury or traumatic brain injury
4. Subjects with a cavity structure that would preclude successful transplantation, as identified on MRI, which may include septations or irregularities in tissue structure
5. Persons with syringomyelia, defined as those with progressively enlarging cysts on T2-weighted images associated with neurological decline
6. Inability to communicate effectively with neurological examiner such that the validity of patient data could be compromised
7. Organ damage or systemic disease that would create an unacceptable risk for surgery or immunosuppression
8. Need for mechanical support of ventilation (ventilator, continuous positive airway pressure [CPAP], bi-level positive airway pressure [BiPAP]), excluding supplemental oxygen, at baseline
9. History of any malignancy (except non-melanoma skin cancers). For cancers in remission for more than five years, enrollment is allowed with concurred documented approval of principal investigator, oncologist, and Sponsor's medical monitor prior to enrollment
10. Pregnant or nursing women
11. Subjects with an implanted spinal cord stimulator (SCS), whether temporary or permanent.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Estimated)
Dates: Start 2025-06-30 (Actual); Primary Completion 2027-08-10 (Estimated); Study Completion 2037-06-30 (Estimated)

PRIMARY OUTCOMES:
Frequency and Severity of Adverse Events Related to the Delivery Device or Injection Procedure Through 30 Days | One month after LCTOPC1 injection
  Frequency and severity of the MI PSD System or injection procedure related adverse events (AEs) through 30 days (1 month).

SECONDARY OUTCOMES:
Frequency and Severity of Adverse Events Related to LCTOPC1 and/or the Concomitant Immunosuppression Through 90 Days | Three months after LCTOPC1 injection
  Frequency and severity of AEs through 90 days (3 months) following injection of LCTOPC1 and/or the concomitant immunosuppression administered.
Incidence of MRI Findings Indicative of Deterioration or Safety-Related Changes at 90 Days | Three months after LCTOPC1 injection
  Incidence of MRI findings indicative of deterioration or safety-related changes at 90 days post-administration of LCTOPC1. Central radiologists will assess MRI data for the presence and severity of: (1) Intramedullary hemorrhage, CSF leak, epidural abscess, or infection; (2) Expanding cyst or mass at the injection site or elsewhere in the CNS; (3) Inflammatory lesions at the injection site or elsewhere in the CNS; (4) CSF flow obstruction. Severity will be categorized as [mild, moderate, severe] based on predefined radiological criteria.

CONTACTS AND LOCATIONS:
Locations (2):
- United States (2):
  - Rancho Research Institue, Downey, California
  - University of California, San Diego, La Jolla, California

IPD SHARING:
Plan to Share IPD: No
At this time, we do not plan to share IPD from this study. As this is a Phase 1 safety study with a small sample size, the data are primarily focused on initial safety assessments and sharing IPD is not anticipated to provide significant additional value. However, summary-level results will be made available in accordance with regulatory guidelines.